CLINICAL TRIAL: NCT04267016
Title: A Clinical Pilot Study to Test the Acceptability and Feasibility of TruGraf® Testing as Part of the Standard of Care
Brief Title: Acceptability and Feasibility of TruGraf® Testing as Part of the Standard of Care
Status: Terminated | Type: Observational
Why Stopped: Sponsor decision to cancel study
Sponsor: Transplant Genomics, Inc. (Industry)
Collaborators: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: TGRP01-US001
Record Dates: First submitted 2020-02-06; First posted 2020-02-12 (Actual); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: Kidney Transplant Rejection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All Subjects Enrolled: Renal transplant recipients who are undergoing routine management
  Interventions: Diagnostic Test: TruGraf Testing - Peripheral blood gene expression profiling

INTERVENTIONS:
Diagnostic Test: TruGraf Testing - Peripheral blood gene expression profiling — 5 mL collection PAXgene blood sample
  Other Names: Standard of care

SUMMARY:
This is an observational study in renal transplant recipients to evaluate the acceptability, feasibility, and clinical utility of TruGraf® testing in conjunction with standard clinical assessment. TruGraf is the first and only non-invasive test approved by Medicare to rule out silent rejection in stable kidney transplant recipients.

ELIGIBILITY:
Inclusion Criteria:

* Recipient of a primary or subsequent deceased-donor or living donor kidney transplantation.
* Stable serum creatinine (current serum creatinine <2.3 mg/dl, <20% increase compared to the average of the previous 3 serum creatinine levels)
* Kidney transplant patients who >90 days (+/- 2 weeks) post-transplant will be included in this study

Exclusion Criteria:

* Need for combined organ transplantation with an extra-renal organ and/or islet cell transplant.
* Recipients of previous non-renal solid organ and/or islet cell transplantation.
* Infection with HIV.
* Infection with BK nephropathy.
* Patients that have nephrotic proteinuria (urine protein >3 gm/day).

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All eligible renal transplant recipients who meet the inclusion/exclusion criteria will be part of this study.
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2020-08-19 (Actual); Primary Completion 2021-05-11 (Actual); Study Completion 2021-05-11 (Actual)

PRIMARY OUTCOMES:
Clinical Utility of TruGraf Results | through study completion, an average of 6 months
  Percent of total number of TruGraf results that the PI identified as having clinical utility
Correlation of TruGraf Results | through study completion, an average of 6 months
  Percent of total number of TruGraf results that the PI identified as being correlated to other clinical results obtained through the standard of care.
Feasibility of TruGraf Testing | through study completion, an average of 6 months
  Percent of total number of eligible subjects for whom the PI was able to complete the entire TruGraf testing workflow

CONTACTS AND LOCATIONS:
Overall Officials: Patty West-Thielke, PharmD, Study Director — Transplant Genomics, Inc.
Locations (1):
- Duke University, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Marsh CL, Kurian SM, Rice JC, Whisenant TC, David J, Rose S, Schieve C, Lee D, Case J, Barrick B, Peddi VR, Mannon RB, Knight R, Maluf D, Mandelbrot D, Patel A, Friedewald JJ, Abecassis MM, First MR. Application of TruGraf v1: A Novel Molecular Biomarker for Managing Kidney Transplant Recipients With Stable Renal Function. Transplant Proc. 2019 Apr;51(3):722-728. doi: 10.1016/j.transproceed.2019.01.054. Epub 2019 Jan 26. PMID 30979456
- [Background] First MR, Peddi VR, Mannon R, Knight R, Marsh CL, Kurian SM, Rice JC, Maluf D, Mandelbrot D, Patel A, David J, Schieve C, Lee D, Lewis P, Friedewald JJ, Abecassis MM, Rose S. Investigator Assessment of the Utility of the TruGraf Molecular Diagnostic Test in Clinical Practice. Transplant Proc. 2019 Apr;51(3):729-733. doi: 10.1016/j.transproceed.2018.10.024. Epub 2018 Dec 11. PMID 30979457